CLINICAL TRIAL: NCT00169949
Title: Open-Label Study of Aripiprazole in Individuals at Risk for Chronic Mental Illness
Brief Title: Aripiprazole Treatment of the Prodrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated due to low enrollment.
Sponsor: Northwell Health (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-134; 03-134
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2009-09-25 (Estimated); Status verified 2007-04

CONDITIONS: Prodromal Schizophrenia; Prodromal Psychosis
Keywords: early intervention; social functioning; role functioning; cognition
MeSH Terms: conditions — Schizotypal Personality Disorder; Social Adjustment | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: aripiprazole

SUMMARY:
The RAP Program is conducting a research study of the antipsychotic medication Aripiprazole. This drug has been approved for treating symptoms associated with schizophrenia and is associated with fewer side effects. This study will explore how well Aripiprazole treats symptoms of early-onset psychotic disorders as well as symptoms that may indicate risk for such disorders, including unusual thoughts, suspiciousness, perceptual abnormalities, social isolation, and sudden changes in functioning.

DETAILED DESCRIPTION:
During the 12-week study, eligible patients are seen 7-9 times by research raters and psychiatrists. These visits include side effect monitoring, scheduled medication increases, and ratings designed to measure subtle improvement of symptoms. Monthly blood and urine samples are collected for safety and substance abuse monitoring, and neuropsychological testing is conducted at the first and last appointments. Participants are compensated for their participation and receive medication and study-related visits at no cost during the trial. Depending on their level of response to the medication, participants may also be eligible for a 3-month extension phase.

ELIGIBILITY:
Inclusion Criteria:

* You are between the ages of 13 and 22.
* You are English-speaking.
* You have a diagnosed psychotic disorder, including: schizophrenia, schizophreniform disorder, schizoaffective disorder, or other psychotic disorder
* OR -
* You are experiencing one or more pre-psychotic symptoms like unusual thoughts, suspiciousness, or unusual perceptual experiences.
* You meet additional RAP criteria assessed during screening and interview.

Exclusion Criteria:

* You have a diagnosis of bipolar disorder or major depression with psychotic features.
* You have a history of neurological, neuroendocrine, or other medical conditions known to affect the brain.
* You have past or current substance dependence.
* You are currently taking Aripiprazole.
* You have taken Aripiprazole in the past.
* You are currently taking and responding well to another medication.

Ages: 13 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30
Dates: Start 2004-01; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Score on attenuated positive symptom scale at 12 weeks
Score on attenuated negative symptom scale at 12 weeks
Score on adverse events rating scale at 12 weeks

SECONDARY OUTCOMES:
Score on social functioning scale at 12 weeks
Score on academic functioning scale at 12 weeks
Score on cognitive measures at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Cornblatt, PhD, Principal Investigator — LIJMC
Locations (1):
- RAP Program, Dept. of Psychiatry Research, The Zucker Hillside Hospital, Glen Oaks, New York, United States